CLINICAL TRIAL: NCT01223768
Title: Acetyl-L-Carnitine In Severe Hepatic Encephalopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Catania (Other)
Other Study IDs: 8-12-00 C
Record Dates: First submitted 2010-10-18; First posted 2010-10-19 (Estimated); Last update posted 2010-10-19 (Estimated); Status verified 2000-12

CONDITIONS: Hepatic Encephalopathy (Grade 3 of the West Haven Grading Scale)
MeSH Terms: conditions — Hepatic Encephalopathy | interventions — Acetylcarnitine

ARMS (2):
- Acetyl-L-carnitine (Experimental)
  Interventions: Drug: Acetyl-l-Carnitine
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Acetyl-l-Carnitine — 2g per day
  Arms: Acetyl-L-carnitine
Drug: placebo — twice per day
  Arms: placebo

SUMMARY:
To assess the clinical efficacy of ALC in the treatment of severe hepatic encephalopathy (grade 3 of the West Haven grading scale), we performed a randomised, double blind placebo-controlled study administering ALC to cirrhotic patients, evaluating the effects on ammonia levels and performance in cognitive functions.

ELIGIBILITY:
Inclusion Criteria:

* patients with severe hepatic encephalopathy (grade 3 of the West Haven grading scale) with hepatic cirrhosis

Exclusion Criteria:

* Patients with a history of recent alcohol abuse, patients using psychotropic drugs (e.g., antipsychotics, interferon, benzodiazepines, anti-epileptics, sedatives and antidepressants)
* Other exclusion criteria were the following: major complications of portal hypertension, such as gastrointestinal blood loss, hepatorenal syndrome or bacterial peritonitis; acute superimposed liver injury;patients with metabolic disorders such as diabetes mellitus, unbalanced heart failure and/or respiratory failure or end-stage renal disease; any additional precipitating factors such as high protein intake (additional high-protein meals), constipation; illiteracy.

Ages: 40 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2002-07; Study Completion 2005-12

CONTACTS AND LOCATIONS:
Locations (1):
- Cannizzaro Hospital, Catania, Italy